CLINICAL TRIAL: NCT06792786
Title: Multi-center Prospective Study of Immunoconsolidation Therapy After Chemoradiotherapy for Esophageal Cancer Based on CtDNA Dynamic Detection
Brief Title: Dynamic Changes of CtDNA to Evaluate the Efficacy of Immunoconsolidation Therapy After Radiotherapy and Chemotherapy for Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Central Hospital of Lishui City (Other)
Collaborators: Jinhua Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Zhifeng Tian,MD, professor, The Central Hospital of Lishui City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZJLSRT002
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer; CtDNA
Keywords: esophageal cancer; radiotherapy; chemotheropy化学疗法; Immunotherapy; ctDNA
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chemoradiotherapy Sequential Toripalimab (Experimental)
  Interventions: Diagnostic Test: ctDNA detection

INTERVENTIONS:
Diagnostic Test: ctDNA detection — dynamically monitor the changes of ctDNA in patients with esophageal cancer Radiation: Radiotherapy 95% PTV50-50.4Gy/25-28fractions, 1.8-2Gy/1 fractions; 5 days a week; 6 weeks. Chemotherapy:weekly paclitaxel (50mg/m²) in combination with carboplatin (AUC=2) chemotherapy, a total of 4-5 cycles.
  Other Names:
  Intensity-modulated radiotherapy (IMRT) Drug: Toripalimab Toripalimab (240 mg, intravenously infused) will be administered as the maintenance treatment every 3 weeks within 4 weeks after the completion of radiotherapy for 1 years or until progression, intolerable toxicity, or physician/patient decision
  Other Names:
  Immunotherapy ctDNA detection: The first tissue and blood ctDNA test (T0) before treatment is based on next generation sequencing (NGS) technology, and ctDNA test is based on tumor- prior analysis informed assays method. Blood ctDNA testing after chemoradiotherapy was performed every 3 months

SUMMARY:
The incidence and mortality of esophageal squamous cell carcinoma are among the highest in China, and most patients are diagnosed in the middle and late stages. Concurrent chemoradiotherapy is the standard treatment for unresectable locally advanced esophageal squamous cell carcinoma. The 5-year formation rate of advanced esophageal cancer is less than 20%. Immunotherapy for advanced esophageal squamous cell carcinoma has definite efficacy and low toxicity, and the results of combined radiotherapy have also been preliminarily reported. Combined immunotherapy after chemoradiotherapy for esophageal cancer is a feasible combination program. But immunotherapy still lacks ideal biomarkers to screen people for advantage. ctDAN status can accurately guide treatment implementation and predict tumor progression. Studies have shown that ctDNA changes are earlier than imaging findings of recurrence or metastasis, and ctNDA detection can sensitively predict tumor progression and prognosis. Therefore, it is necessary to dynamically monitor the changes of ctDNA in immunoconsolidation therapy after radical radiotherapy and chemotherapy for esophageal cancer, and explore its correlation with the curative effect and prognosis of radical radiotherapy and chemotherapy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

-1. Age 18-75 years old, male or female; 2.ECOG score 0 ~ 1; 3. Esophageal squamous cell carcinoma was confirmed by pathology. 4. No radiotherapy, chemotherapy or other treatment was given before enrollment; 5. AJCC 8th stage II-IVa, which cannot be treated by surgical evaluation or patients reject operation; 6. Has sufficient organ function, (1) Blood routine: Peripheral blood white blood cell count ≥3.0×10^9 / L, neutrophil absolute value ≥1.5×10^9 /L, hemoglobin ≥90 g/L, platelets ≥75×10^9 / L (No blood transfusion and blood products within 14 days, no use of G-CSF and other blood-stimulating factors to correct), (2) Liver function: total bilirubin ≤1.5× upper limit of normal(ULN), AST and ALT≤2.5× ULN, alkaline phosphatase ≤5× ULN, (3) Renal function: Serum creatinine ≤1.0× ULN or crcl ≥50 ml/min, (4) Adequate haemostasis laboratory data prior to randomization: INR or PT ≤1.5×ULN (If the subject was receiving anticoagulant therapy, as long as the PT was within the intended use range of anticoagulant drugs) (5) Myocardial enzymes were within the normal range.

7. Sign a consent form.

Exclusion Criteria:

* 1. unable to provide a sufficient number of tissue samples/blood samples for the study prior to treatment; 2. The patient refused to accept dynamic ctDNA testing; 3. A history of malignant tumors other than esophageal cancer in the past 5 years (excluding cured local tumors such as cervical carcinoma in situ, basal cell carcinoma, and prostate carcinoma in situ); 4. A history of gastrointestinal bleeding within the past 6 months, or abnormal coagulation at enrollment, or currently receiving thrombolytic or anticoagulant therapy, indicating a higher risk of bleeding; 5. Severe cardiovascular and cerebrovascular diseases; 6. History of interstitial lung disease or active pneumonia/tuberculosis; 7. Severe allergic reaction to paclitaxel/cisplatin chemotherapeutics or any monoclonal antibody; 8. Other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | two years
  We aim to evaluate the progression-free survival (PFS) of patients with unresectable esophageal squamous cell carcinoma who accept concurrent chemoradiotherapy and received sequential treatment with Triptolide injection after radiotherapy.

SECONDARY OUTCOMES:
locoregional progression-free survival (LRPFS) | 2 years
  locoregional progression-free survival (LRPFS) is defined as the time from treatment to the primary tumor or regional lymph node histopathological progressconfirmed on CT. In the absence of pathology, tumor progression is evident under gastroscopy and/or confirmed by imaging such as PET-CT.
Overall survival (OS) | 2 years
  Overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - The central Hospital of Lishui City, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
The results of the study were inconclusive.